CLINICAL TRIAL: NCT03436160
Title: Exploratory Microdose Study Assessing Pharmacokinetics and Bioavailability of Three Novel Triazine Compounds
Brief Title: Study Assessing Pharmacokinetics and Bioavailability of Three Novel Triazine Compounds
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-15-45
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of three groups to receive 100 mcg Carbon-14 radio labeled WR826647, WR909388, or WR909390
Masking Description: Blinding is not necessary in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- WR826647 (Experimental): 100 mcg Carbon-14 radio labeled WR826647 administered via IV
  Interventions: Drug: WR826647
- WR909388 (Experimental): 100 mcg Carbon-14 radio labeled WR909388 administered via IV
  Interventions: Drug: WR909388
- WR909390 (Experimental): 100 mcg Carbon-14 radio labeled WR909390 administered via IV
  Interventions: Drug: WR909390

INTERVENTIONS:
Drug: WR826647 — 100 mcg Carbon-14 radio labeled WR826647 at an exposure no greater than 250 nCi per dose, administered both IV (bolus) and PO with a six half-life wash-out period between IV and PO administration. Interim analyses will be done at Day 14 following the IV dosing groups in order to assess half-lives of the three compounds to ensure the wash-out period between IV and PO dosing is at least six half-lives long.
  Other Names: Triazine WR826647
  Arms: WR826647
Drug: WR909388 — 100 mcg Carbon-14 radio labeled WR909388 at an exposure no greater than 250 nCi per dose, administered both IV (bolus) and PO with a six half-life wash-out period between IV and PO administration. Interim analyses will be done at Day 14 following the IV dosing groups in order to assess half-lives of the three compounds to ensure the wash-out period between IV and PO dosing is at least six half-lives long.
  Other Names: Triazine WR909388
  Arms: WR909388
Drug: WR909390 — 100 mcg Carbon-14 radio labeled WR909309 at an exposure no greater than 250 nCi per dose, administered both IV (bolus) and PO with a six half-life wash-out period between IV and PO administration. Interim analyses will be done at Day 14 following the IV dosing groups in order to assess half-lives of the three compounds to ensure the wash-out period between IV and PO dosing is at least six half-lives long.
  Other Names: Triazine WR909390
  Arms: WR909390

SUMMARY:
Open-label, randomized, microdose study

DETAILED DESCRIPTION:
This is an open-label, randomized, fixed-sequence, microdose study of three Carbon-14 radio labeled (14C) triazine compounds WR826647, WR909388, WR909390 designed in accordance with ICH Guidance for Industry M3(R2) (ICH 2009). Subjects will be randomized to one of three groups to receive 100 mcg WR826647, WR909388, or WR909390 at an exposure no greater than 250 nCi per dose, administered both IV (bolus) and PO with a six half-life wash-out period between IV and PO administration. Interim analyses will be done at Day 14 following the IV dosing groups in order to assess half-lives of the three compounds to ensure the wash-out period between IV and PO dosing is at least six half-lives long.

Pharmacokinetic parameters of the 3 compounds will be calculated from the plasma-time data using Phoenix WinNonlin version 6.3 or higher, and descriptive statistics assessed using SAS version 9.3 or higher. No statistical significance inferences will be made. An analysis of variance (ANOVA) will be performed on the natural logarithm (ln) transformed dose-adjusted AUCinf to estimate the bioavailability. The sample size of 6 subjects per group is considered adequate to obtain useful data to compute descriptive statistics. Interim analyses will be done after the IV dosing groups in order to assess half-lives of the 3 compounds to ensure the wash-out period between IV bolus and oral dosing is at least 6 half-lives long.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-breastfeeding female of non-childbearing potential (defined as either surgically sterilized by bilateral tubal ligation or hysterectomy with bilateral ophorectomy at least 6 months before dosing, or is one year post-menopausal, confirmed by screening follicle-stimulating hormone [FSH] serum levels consistent with postmenopausal status >30mIU/mL)
* Between the ages of 19 and 50, inclusive, at the time of screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or EKGs, as deemed by the PI or designee.
* Body Mass Index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2 at screening.
* Continuous non smoker who has not used nicotine containing products for at least 90 days prior to the first dose and throughout the study.
* A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to first dose/dosing of study drug. A male who has been vasectomized less than 4 months prior to study first dose/dosing must follow the same restrictions as a non vasectomized male).
* Male volunteers must agree not to donate sperm from the first dose until 90 days after last dose.
* Ability to comprehend and willingness to sign informed consent, which includes the Authorization for the Release of Health Information document
* Willingness to comply with all study procedures including two 24-hour inpatient stays at the study clinic and returning to the clinic for scheduled follow-up visits

Exclusion Criteria:

* History of any medical or psychiatric illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds (i.e., compound in the same family).
* Positive urine drug results for alcohol, amphetamines, methamphetamines, cocaine, or opioids at screening or first check in.
* Positive results at screening for HIV, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Received any other investigational drug within 30 days prior to study entry. The 30 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.
* An employee of the study site involved with the study
* Inability to comply with the study procedures
* Unable to refrain from or anticipate the use of any drug, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dose and throughout the study. Acetaminophen (up to 2 g per 24 hour period may be permitted during the study but only for dosing as needed to treat adverse events (AEs).
* Unable to refrain from or anticipate the use of any drugs known to be significant inducers of cytochrome P450 (CYP) enzymes and/or permeability glycoprotein (P gp), including St. John's Wort, for 30 days prior to the first dose/dosing and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/pharmacodynamics interaction with study drug.
* Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 30 days prior to the first dose and throughout the study.
* Donation of blood or significant blood loss within 56 days prior to the first dose.
* Plasma donation within 7 days prior to the first dose.
* Subjects with tattoo(s) or scarring at or near the site of IV infusion or any other condition which may interfere with infusion site examination(s), in the opinion of the Investigator or designee.
* Participation in another clinical trial in which a 14C-labeled drug was administered within 1 year prior to Day 1.
* Any other significant finding that in the opinion of the clinical investigators would make the subject's participation in the study unsafe.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2018-11-03 (Actual); Study Completion 2018-11-03 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic parameters of Carbon-14 radio labeled (14C) WR826647, WR909388, and WR909390 | 0, 5, 15 min, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours, and then daily for 1 week, and weekly until 3 weeks following dosing
  Pharmacokinetic parameters of the 3 compounds will be calculated from the plasma-time data and descriptive statistics assessed . No statistical significance inferences will be made.

SECONDARY OUTCOMES:
Bioavailability of Carbon-14 radio labeled (14C) WR826647, WR909388, and WR909390 | 0, 5 , 15 min, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours, and then daily for 1 week, and weekly until 3 weeks following dosing.
  An analysis of variance (ANOVA) will be performed on the natural logarithm (ln) transformed dose-adjusted AUCinf to estimate the bioavailability.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Hunt, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided